CLINICAL TRIAL: NCT04758390
Title: Multilevel Comprehensive HIV Prevention Package for South African Adolescent Girls and Young Women
Brief Title: A Comprehensive HIV Prevention Package for South African Adolescent Girls and Young Women
Acronym: IMARA-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Desmond Tutu Health Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Natasha Crooks, Assistant Professor, Human Development Nursing Science, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-0709; UH3HD096875 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Sexually Transmitted Infections; HIV Infections
Keywords: HIV prevention; Adolescent girls and young women; South Africa; Mother-daughter intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections

STUDY DESIGN:
Intervention Model Description: Adolescent girl and young women-female caregiver (AGYW-FC) dyads will be randomized to the IMARA intervention arm or a health promotion control arm matched in time and intensity. IMARA and the health promotion program will be delivered as group interventions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMARA intervention arm (Experimental): Participants randomized to the IMARA arm will receive the IMARA intervention (i.e., the intervention group).
  Interventions: Behavioral: IMARA (intervention group)
- Health promotion control arm (Experimental): Participants randomized to the health promotion control arm will receive the health promotion intervention (i.e., the control group).
  Interventions: Behavioral: Health promotion control group

INTERVENTIONS:
Behavioral: IMARA (intervention group) — The IMARA intervention aligns with an ecological framework, emphasizing the intersection of individual, social, and structural determinants of women's sexual health and behavior. Separate FC and AGYW groups run simultaneously and cover parallel content, while joint activities enhance FC credibility as a resource for HIV/STI prevention and facilitate practice of communication skills. Interventionists use interactive and experiential activities. IMARA's goals and motto emphasize strong FC-AGYW relationships, sisterhood, community empowerment, and motivation for HIV prevention, and build group cohesion. FC and AGYW sign a pact to confirm commitment to the program. At the end of Workshop Day 1, participants receive homework to complete during the week. Woven throughout IMARA is the impact of mental health issues, alcohol and drug use, and violence on HIV-risk.
  Arms: IMARA intervention arm
Behavioral: Health promotion control group — The health promotion control intervention is a family-based intervention previously delivered to families in SA and translated into isiXhosa. The intervention promotes healthy living by encouraging good nutrition, exercise, and violence reduction. It will be delivered in the same format as IMARA and will be identical in length and intensity.
  Arms: Health promotion control arm

SUMMARY:
To achieve an AIDS-free generation, there is a critical need for programs which go beyond individual-level behavior change to reduce HIV and STI infections among adolescent girls and young women in sub-Saharan Africa. Informed, Motivated, Aware, and Responsible Adolescents and Adults (IMARA) is an evidence-based HIV-prevention intervention for adolescent girls and young women (AGYW) and their female caregivers, which has been adapted for a South African audience. The study will test whether AGYW receiving IMARA will have fewer sexually-transmitted infections (STI) and greater acceptance of HIV testing and counseling (HTC) and pre-exposure prophylaxis (PrEP) at 6-month follow-up compared to AGYW assigned to the health-promotion control intervention.

DETAILED DESCRIPTION:
Reducing new HIV and STI infections among South African (SA) adolescent girls and young women (AGYW) is global public health priority. SA has the world's largest HIV epidemic, and SA AGYW acquire HIV at twice the rate of and seroconvert on average 5 - 7 years earlier than male peers. As new infections continue to outpace access to and availability of pre-exposure prophylaxis (PrEP) and antiretroviral therapy (ART), primary prevention remains the most viable strategy to stem new transmission. SA efforts to prevent HIV transmission in youth focus mostly on individual-level behavior change, but AGYW's persistent HIV disparities are explained by broad social and structural inequities that shape and constrain HIV-risk behaviors. Comprehensive HIV prevention packages that are integrated, synergistic, and tailored to the local epidemiology and cultural context are likely to achieve and sustain maximum reductions in HIV-risk. Female caregivers (FC) are an untapped resource in the HIV prevention toolbox and offer a novel opportunity to strengthen AGYW prevention efforts. AGYW may also be change agents for their FC who want to be positive role models for AGYW, and thus, adopt HIV prevention behaviors, including HTC and PrEP.

This study will evaluate the effectiveness and cost-effectiveness of Informed Motivated Aware and Responsible Adolescents and Adults (IMARA), a multilevel, innovative, family-based HIV prevention program that targets individual, social, and structural drivers of risk. IMARA demonstrated a 43% reduction in incident STI at 12-month follow-up among black 14-18-year-old girls in the US. IMARA has been systematically tailored for the SA context and piloted among AGYW and FC dyads. A two-arm RCT will now be conducted with about 645 AGYW (15-19 years old) and FC dyads. Following randomization, AGYW-FC dyads will participate in a 2-day group workshop (~12 hours) that includes joint and separate mother and daughter activities. AGYW and FC will complete baseline, 6-, and 12-month assessments, including testing for three STI (chlamydia, gonorrhea, and trichomoniasis). We will offer HTC and PrEP at each assessment and track uptake and linkage to care. AGYW and FC who are HIV-negative and interested in PrEP will receive a one-month supply and referral to a clinic. They will additionally receive treatment and counseling if testing positive for an STI and referral for care at an ART clinic if testing positive for HIV. Data will be collected to determine the costs of IMARA. Analyses will compare AGYW across the intervention and control programs on STI incidence, and PrEP and HTC uptake, in addition to secondary outcomes. We will also evaluate the costs and cost-effectiveness of IMARA with respect to the acquisition of STI and HIV, where possible considering power limitations. Additionally, the intervention's implementation will be explored. The study answers an urgent need to evaluate the effectiveness and cost-effectiveness of combination HIV prevention packages for AGYW.

ELIGIBILITY:
Inclusion criteria for AGYW include:

* female;
* 15-19 years-old;
* residing in Klipfontein/Mitchells Plain (K/MP);
* speak isiXhosa or English or a combination of these languages;
* willing to have biometric data collected.

Inclusion criteria for FC include:

* identified by AGYW as a FC;
* 24 years and older;
* living with or in daily contact with the AGYW;
* speak isiXhosa or English or a combination of these languages;
* willing to have biometric data collected.

Exclusion Criteria:

* AGYW will be excluded from the study if they do not have a FC to participate in the study.
* AGYW and FC will be excluded from the study if they are: a) unable to understand the consent/assent process and provide written informed consent; b) currently enrolled in another research study addressing HIV/STIs/PrEP.
* AGYW and FC must agree to participate as a dyad. AGYW refusal will supersede FC consent.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants will be eligible to participate if they are female.
Enrollment: 1290 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Proportion of adolescent girls and young women (AGYW) with a sexually-transmitted infection (STI) at baseline and midline | ~6 months (from baseline to midline)
  A positive test for at least one of three STIs: chlamydia, gonorrhea, and/or trichomoniasis
Proportion of AGYW who complete HIV testing and counseling (HTC) at baseline and midline | ~6 months (from baseline to midline)
  Completion of HTC
Proportion of AGYW who elect to take pre-exposure prophylaxis (PrEP) at baseline and midline | ~6 months (from baseline to midline)
  Uptake of PrEP

SECONDARY OUTCOMES:
Proportion of AGYW with an STI at baseline and endline | ~12 months (from baseline to endline)
  A positive test for at least one of three STIs: chlamydia, gonorrhea, and/or trichomoniasis
Proportion of AGYW who complete HTC at baseline and endline | ~12 months (from baseline to endline)
  Completion of HTC
Proportion of AGYW who elect to take PrEP at baseline and endline | ~12 months (from baseline to endline)
  Uptake of PrEP
Proportion of AGYW who report risky sexual behavior at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  Sexual behavior (e.g., condom use, substance use during sex, number of partners, concurrent partners) will be measured via self-report using the AIDS Risk Behavior Assessment (ARBA) (Donenberg, 2001).
Proportion of AGYW who report adherence to PrEP at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  Adherence to PrEP (where appropriate) will be measured via self-report using items from the Wilson scale (2017)
Proportion of AGYW who report adherence to antiretroviral therapy (ART) at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  Adherence to ART (where appropriate) will be measured via self-report using items from the Wilson scale (2017)
Proportion of AGYW who test positive for HIV at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  A positive test for HIV during HTC
Intervention cost-effectiveness | The study duration (~2.5 years)
  The cost-effectiveness ratio, defined as the incremental cost of the IMARA intervention per infection prevented by the intervention.

OTHER OUTCOMES:
Proportion of female caregivers (FC) with an STI at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  A positive test for at least one of three STIs: chlamydia, gonorrhea, and/or trichomoniasis
Proportion of FC who complete HTC at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  Completion of HTC
Proportion of FC who elect to take PrEP baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  Uptake of PrEP
Proportion of FC who report risky sexual behavior at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  Sexual behavior (e.g., condom use, substance use during sex, number of partners, concurrent partners) will be measured via self-report using the AIDS Risk Behavior Assessment (ARBA) (Donenberg, 2001)
Proportion of FC who test positive for HIV at baseline, midline, and endline | ~6 months (from baseline to midline) and ~12 months (from baseline to endline)
  A positive test for HIV during HTC
Intervention feasibility | The study duration (~2.5 years)
  Feasibility will be measured through surveys completed by participants and study staff using items adapted from the Johns Hopkins' Applied Mental Health Research (AMHR) implementation science measure (Haroz et al, 2019).
Intervention acceptability | The study duration (~2.5 years)
  Acceptability will be measured through surveys completed by participants and study staff using items adapted from the Johns Hopkins' AMHR implementation science measure (Haroz et al, 2019).
Intervention appropriateness | The study duration (~2.5 years)
  Appropriateness will be measured through surveys completed by participants and study staff using items adapted from the Johns Hopkins' AMHR implementation science measure (Haroz et al, 2019).
Intervention reach | The study duration (~2.5 years)
  Reach will be assessed through surveys completed by participants and study staff using items adapted from the Johns Hopkins' AMHR implementation science measure (Haroz et al, 2019).
Intervention adoption | The study duration (~2.5 years)
  Adoption will be assessed through surveys completed by participants and study staff using items adapted from the Antiretroviral Treatment Access Study (ARTAS) (Norton et al, 2012).
Intervention fidelity | The study duration (~2.5 years)
  Fidelity will be assessed by facilitators and observers of the intervention using an adapted version of the Treatment Fidelity Questionnaire (Lane et al, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Geri R Donenberg, PhD, Principal Investigator — University of Illinois at Chicago; Linda-Gail Bekker, MBChB, PhD, Principal Investigator — Desmond Tutu Health Foundation
Locations (1):
- Desmond Tutu Health Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be placed in one or more electronic databases (e.g. DASH, PATC3H) which could be used for other research studies in addition to this one.
Supporting Information: Study Protocol
Time Frame: Data sharing will generally coincide with publication of the study's main findings no later than 1 year after acceptance of the primary manuscript or study closure, whichever comes first.
Access Criteria: To access data in the DASH repository, users will be required to register in DASH, belong to an institution with an approved assurance from the Department of Health and Human Services Office for Human Research Protections, submit a research plan, execute a DASH data use agreement, submit approval from their local IRB, obtain approval by the DASH Data Access Committee, and obtain approval from the Study-Specific Approving Entity. To access data through the PATC3H consortium, researchers must be on one of the PATC3H consortium research teams; the decision to share data will be at the discretion of the principal investigator.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] Donenberg GR, Kendall AD, Emerson E, Fletcher FE, Bray BC, McCabe K. IMARA: A mother-daughter group randomized controlled trial to reduce sexually transmitted infections in Black/African-American adolescents. PLoS One. 2020 Nov 2;15(11):e0239650. doi: 10.1371/journal.pone.0239650. eCollection 2020. PMID 33137103
- [Background] Atujuna M, Merrill K, Ndwayana S, Emerson E, Fynn L, Bekker L-G, Donenberg G: Engaging female caregivers to improve South African girls' and young womens' sexual and reproductive health outcomes. In: HIV Research for Prevention Virtual Conference. 2021.
- [Background] Donenberg GR, Emerson E, Bryant FB, Wilson H, Weber-Shifrin E. Understanding AIDS-risk behavior among adolescents in psychiatric care: links to psychopathology and peer relationships. J Am Acad Child Adolesc Psychiatry. 2001 Jun;40(6):642-53. doi: 10.1097/00004583-200106000-00008. PMID 11392341
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Background] Haroz EE, Bolton P, Nguyen AJ, Lee C, Bogdanov S, Bass J, Singh NS, Doty B, Murray L. Measuring implementation in global mental health: validation of a pragmatic implementation science measure in eastern Ukraine using an experimental vignette design. BMC Health Serv Res. 2019 Apr 29;19(1):262. doi: 10.1186/s12913-019-4097-y. PMID 31036002
- [Background] Lane KL, Bocian KM, MacMillan DL, Gresham FM. Treatment integrity: An essential-but often forgotten-component of school-based interventions. Preventing School Failure. 2004; 48(3): 36-43.
- [Background] Norton WE. An exploratory study to examine intentions to adopt an evidence-based HIV linkage-to-care intervention among state health department AIDS directors in the United States. Implement Sci. 2012 Apr 2;7:27. doi: 10.1186/1748-5908-7-27. PMID 22471965
- [Derived] Donenberg G, Merrill KG, Atujuna M, Emerson E, Bray B, Bekker LG. Mental health outcomes of a pilot 2-arm randomized controlled trial of a HIV-prevention program for South African adolescent girls and young women and their female caregivers. BMC Public Health. 2021 Nov 30;21(1):2189. doi: 10.1186/s12889-021-12010-1. PMID 34847908
- [Derived] Donenberg GR, Atujuna M, Merrill KG, Emerson E, Ndwayana S, Blachman-Demner D, Bekker LG. An individually randomized controlled trial of a mother-daughter HIV/STI prevention program for adolescent girls and young women in South Africa: IMARA-SA study protocol. BMC Public Health. 2021 Sep 20;21(1):1708. doi: 10.1186/s12889-021-11727-3. PMID 34544403